CLINICAL TRIAL: NCT01585389
Title: Expression and Subcellular Localization of NEIL3 in Tumors
Brief Title: Studying Gene Expression and Location in Samples From Patients With Brain Tumors
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ABTR12B3; COG-ABTR12B3 (Other: Children's Oncology Group); ABTR12B3 (Other: Children's Oncology Group); CDR0000732178 (Other: Clinical Trials.gov); NCI-2012-00731 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult brain tumor; childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Gene Expression Profiling; Genetic Linkage; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: genetic linkage analysis
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to brain tumors.

PURPOSE: This research studies gene expression and location in samples from patients with brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the expression and subcellular localization of nei endonuclease VIII-like 3 (NEIL3) in brain tumors.

OUTLINE: Tissue microarray samples are analyzed for NEIL3 expression and subcellular localization by immunohistochemical methods.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tissue microarrays (TMA) samples from the Biopathology Core
* Samples from patients diagnosed with brain tumors

  * Progenitor, or blast, cell origin

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with brain tumors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Correlation of NEIL3 expression and/or nuclear localization with tumor type or grade with respect to degree of differentiation

CONTACTS AND LOCATIONS:
Overall Officials: Heithem M. El-Hodiri, PhD, Principal Investigator — Nationwide Children's Hospital